CLINICAL TRIAL: NCT03923257
Title: Phase I Trial of Peptide Receptor Radiotherapy (PRRT) With 177Lu-DOTA-tyr3-Octreotate (177Lu-DOTATATE) in Children and Adolescents With Neuroendocrine Tumor or Pheochromocytoma/Paraganglioma
Brief Title: Dosimetry Guided PRRT With 177Lu-DOTATATE in Children and Adolescents
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: competing clinical trial opening
Sponsor: Sue O'Dorisio (Other)
Collaborators: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor-Investigator, Sue O'Dorisio, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201812772
Record Dates: First submitted 2019-03-29; First posted 2019-04-22 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Neuroendocrine Tumors; Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Neuroendocrine Tumors; Pheochromocytoma; Paraganglioma | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRRT with 177Lu-DOTA-tyr3-OCTREOTATE (Experimental): 177Lu-DOTA-tyr3-OCTREOTATE (177Lu-DOTATATE) and amino acid will be administered intravenously (IV) on Day 1 of each of four treatment cycles, 8 weeks apart.
  This study will consist of children and adolescents ages 1-20 years with relapsed or refractory neuroendocrine tumors and pheochromocytoma or paraganglioma. Children and adolescents with neuroendocrine tumor, pheochromocytoma or paraganglioma will not have had any previous endoradiotherapy with 90Y-DOTATOC, 131I-MIBG, or 177Lu-DOTATATE.
  Interventions: Drug: 177Lu-DOTA-tyr3-OCTREOTATE; Procedure: Peptide Receptor Radiotherapy (PRRT)

INTERVENTIONS:
Drug: 177Lu-DOTA-tyr3-OCTREOTATE — This is a peptide receptor radiotherapy that targets somatostatin receptors on tumor cells.
  Other Names: Lutathera
Procedure: Peptide Receptor Radiotherapy (PRRT) — PRRT is internal radiation that is individually dosed according to patient body surface area, kidney function and bone marrow status.

SUMMARY:
This is a Phase I/II peptide receptor radiotherapy (PRRT) trial of 177Lu-DOTA-OCTREOTATE in children and adolescents with neuroendocrine tumors and pheochromocytoma or paraganglioma.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to determine if peptide receptor radiotherapy (PRRT) using 177Lu-DOTA-OCTREOTATE given intravenously in children and adolescents is an effective treatment and to describe its toxicities.

This study will consists of children and adolescents ages 1-20 years with relapsed or refractory neuroendocrine tumors and pheochromocytoma or paraganglioma.

ELIGIBILITY:
Inclusion Criteria:

* Disease not amenable to standard treatment (nonresectable or disease present after one or more surgeries and/or Sandostatin treatment) or subject has failed existing first line chemotherapy, biologic therapy, targeted agent therapy or radiation therapy.
* Participation in Iowa Neuroendocrine Tumor Registry and recommendation by University of Iowa PRRT tumor board.
* A pathologically confirmed (histology or cytology) Neuroendocrine Tumor (NET), Pheochromocytoma (PCC), or Paraganglioma (PGL).
* For patients with measurable or evaluable disease: >50% of lesions must demonstrate 68Ga-DOTATATE /DOTATOC uptake greater than physiologic liver uptake by visual assessment. At least one lesion must be confirmed by conventional imaging (CT or MRI).
* For patients with measurable disease, the target lesion is one that either has never received external beam radiation or has been previously irradiated and has since demonstrated progression.
* For patients with no measurable disease (no meaurable target lesions), who have evaluable disease (bone disease, MIBG positive disease, liver metastases not detectable on MRI or CT), the disease must be seen on 68Ga-DOTATATE/DOTATOC PET/CT.
* No previous endogenous radiation with 177Lu-DOTATATE/TOC or 90Y-DOTATATE/TOC or 131I-MIBG within 12 months of most recent treatment.
* Age ≥ 18 months < 20 years at the time of first study drug administration.
* Performance status as determined by Karnofsky ≥ 60 or Lansky Play Scale ≥ 60 at the time of study drug administration.

NOTE: Neurologic deficits in patients with brain metastases must have been stable for at least 7 days prior to study enrollment.

* Completion of validated Pediatric Quality of Life Questionnaire.
* Within seven (7) days of study drug administration, must have normal organ and bone marrow function as defined below:

Adequate Bone Marrow Function Defined as:

* Peripheral absolute neutrophil count (ANC) ≥ 1000/m3
* Platelet count ≥ 75,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Hemoglobin ≥ 8g/dL Organ Function Requirements
* AST(SGOT)& ALT(SGPT) <10X institutional upper limit of normal for age
* Total bilirubin <3X ULN for age
* BUN < 2X normal
* creatinine, Normal for age
* Glomerular filtration rate (GFR) only if creatinine > normal for age
* Nuclear GFR or CrCl ≥ 80 ml/min/1.73m2
* Urinalysis No greater than 1+ hematuria or proteinuria
* The effects of 177Lu-DOTATATE on the developing human fetus are unknown. For this reason and because Class C agents are known to be teratogenic, all subjects capable of becoming pregnant must agree to practice a medically acceptable birth control measure (abstinence, birth control pills, intrauterine devices, vaginal diaphragm, vaginal sponge, or condom with spermicidal jelly) throughout the study and for eight months following the end of the last treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Parent's ability to understand and the willingness to sign a written informed consent document for children < seven (7) years of age. Children ≥ seven (7) years of age will sign assent along with parental consent or will co-sign consent with parent in accordance with rules of the state in which treatment is received.

Exclusion Criteria:

* Pregnant women are excluded from this study because 177Lu-DOTATATE is a Class C agent with potential teratogenic or abortifacient effects.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 177Lu-DOTATATE, breastfeeding should be discontinued until 3 months after the last administration of study drug.
* Major surgery within 8 weeks of study drug administration.
* External beam radiation to both kidneys (scatter doses of <500 cGy to a single kidney or radiation to < 50% of a single kidney is acceptable).
* Prior PRRT with 90Y-DOTATOC (TATE) or 177Lu-DOTATOC (TATE) or 131I-MIBG for this malignancy within 12 months of first study dose.
* Another investigational drug within 8 weeks of study drug administration.
* Concurrent, malignant disease for which patient is on active therapy.
* Another significant medical, psychiatric, or surgical condition which is currently uncontrolled by treatment and which would likely affect the subject's ability to complete this protocol.
* Subjects who have received Sandostatin LAR or long-acting lanreotide in the past 28 days must be appropriately delayed. Subjects may be maintained on short acting octreotide during the time from last injection of long-acting somatostatin analogue until 8-24 hrs prior to injection of study drug.
* Known antibodies to Octreotide, Lanreotide, or DOTATATE or history of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-DOTATATE.
* Uncontrolled illness including, but not limited to ongoing or active infection, uncontrolled diabetes mellitus, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hepatic cirrhosis or severe impairment, or psychiatric illness/social situations that would limit compliance with study requirements.
* Corticosteroids: Patients receiving corticosterods who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, ≥ 14 days must have elapsed since last dose of corticosteroid
* Patients who have received a prior solid organ transplantation are not eligible
* Patients will be excluded if they have a known allergy to any of the drugs used in the study
* Prior Therapy:
* Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive. At least 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea).
* Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or ANC counts): ≥ 7 days after the last dose of agent. Short-acting somatostatin analogue may be administered up to eight hours prior to infusion of study drug.
* Antibodies: ≥ 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to Grade ≤ 1.
* Hematopoietic growth factors: ≥ 14 days after the last dose of a long-acting growth factor (e.g. Peg-Filgrastim) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator.
* Interleukins, Interferons and Cytokines (other than Hematopoietic Growth Factors): ≥ 21 days after the completion of interleukins, interferon or cytokines (other than Hematopoietic Growth Factors).
* Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion or boost infusion: ≥ 84 days after stem cell infusion
* Evidence of GVHD.
* Autologous stem cell infusion including boost infusion: ≥ 42 days; cellular therapy: ≥ 42 days after the completion of any type of cellular therapy (e.g. modified T cells, NK cells, dendritic cells, etc.).

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Toxicities | Initiation of treatment through 5 years
  To examine the toxicity related to the therapy by measuring the number of treatment related adverse events in patients
  Adverse events will be reported in tabular form by type and grade. Adverse events will be graded according to the most recent CTE guidelines.
Objective Response Rate (ORR) according to RECIST criteria in children | Initiation of treatment through 5 years
  To determine overall response rate (ORR) (complete response [CR] + partial response [PR]) + stable disease [SD] per RECIST v1.1)

SECONDARY OUTCOMES:
Measure and demonstrate accuracy of radiation dose to kidneys in children based on a single SPECT/CT image of the kidneys plus a single whole body scan | Initiation of treatment through treatment #4 (approximately 26 weeks)
  Six subjects will have whole body imaging and SPECT/CT of kidneys performed at 3-8 hours plus whole body and SPECT at 20-28 hours, 44-52 hours, 92-100 hours and 116-124 hours after the administration of the radiopharmaceutical. Data will be analyzed using method of Madsen[1,2]. Single point dosimetry will be utilized with subsequent cohorts if data demonstrates agreement with adult dosimetry. Biological effective dose (BED) to kidneys will be calculated according to Bodei et al [3].
  The information on renal uptake, renal mass and residence time will be entered into OLINDA software to calculate the radiation dose. If single point dosimetry proves to be accurate, any remaining Phase I subjects and all Phase II subjects will receive single point dosimetry for both renal and bone marrow radiation dose estimation.
Measure and demonstrate accuracy of radiation dose to bone marrow in children based on radioactivity in a single blood sample | Initiation of treatment through treatment #4 (approximately 26 weeks)
  Blood dosimetry will be performed as a surrogate of bone marrow dosimetry. Blood samples (1 mL) will be obtained prior to start of amino acid infusion and subsequently in the same time frame with the imaging sessions.
Progression Free Survival (PFS) according to RECIST criteria in children | Initiation of treatment through 5 years
  Progression will be defined using the RECIST 1.1 guidelines. Results are provided in nominal categories (CR, PR, SD, PD) as per RECIST.
Measure effect of PRRT in quality of life with the PROMIS Pediatric Profile v2.0 - Profile-37 | Initiation of treatment through treatment #4 (approximately 26 weeks)
  Parents of participants will be asked to complete the PROMIS Pediatric Profile v2.0 - Profile-37

CONTACTS AND LOCATIONS:
Overall Officials: M. Sue O'Dorisio, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madsen MT, Menda Y, O'Dorisio TM, O'Dorisio MS. Technical Note: Single time point dose estimate for exponential clearance. Med Phys. 2018 May;45(5):2318-2324. doi: 10.1002/mp.12886. Epub 2018 Apr 16. PMID 29577338
- [Background] Menda Y, Madsen MT, O'Dorisio TM, Sunderland JJ, Watkins GL, Dillon JS, Mott SL, Schultz MK, Zamba GKD, Bushnell DL, O'Dorisio MS. 90Y-DOTATOC Dosimetry-Based Personalized Peptide Receptor Radionuclide Therapy. J Nucl Med. 2018 Nov;59(11):1692-1698. doi: 10.2967/jnumed.117.202903. Epub 2018 Mar 9. PMID 29523629
- [Background] Bodei L, Cremonesi M, Ferrari M, Pacifici M, Grana CM, Bartolomei M, Baio SM, Sansovini M, Paganelli G. Long-term evaluation of renal toxicity after peptide receptor radionuclide therapy with 90Y-DOTATOC and 177Lu-DOTATATE: the role of associated risk factors. Eur J Nucl Med Mol Imaging. 2008 Oct;35(10):1847-56. doi: 10.1007/s00259-008-0778-1. Epub 2008 Apr 22. PMID 18427807